CLINICAL TRIAL: NCT02245191
Title: Ephedrine, Phenylephrine and Metaraminol Effects on Maternal Cardiac Output, Uterine Blood Flow and Fetal Circulation in Patients With Preeclampsia Under Spinal Anesthesia for Cesarean
Brief Title: Ephedrine, Phenylephrine and Metaraminol Effects on Maternal Cardiac Output, Uterine Blood Flow and Fetal Circulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: VASPRES-3
Record Dates: First submitted 2014-08-07; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-05

CONDITIONS: Preeclampsia
Keywords: Vasopressor; Cesarian delivery; Hypotension; Maternal cardiac output; Uteroplacental blood flow; Cerebral fetal blood flow; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Hypotension | interventions — Ephedrine; Phenylephrine; Metaraminol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ephedrine Group (Experimental): Patients who will receive ephedrine after spinal anesthesia
  Interventions: Drug: Ephedrine
- Phenylephrine Group (Experimental): Patients who will receive Phenylephrine after spinal anesthesia
  Interventions: Drug: Phenylephrine
- Metaraminol (Experimental): Patients who will receive Metaraminol after spinal anesthesia
  Interventions: Drug: Metaraminol

INTERVENTIONS:
Drug: Ephedrine — 5mg after Spinal Anesthesia
  Arms: Ephedrine Group
Drug: Phenylephrine — 100mcg after Spinal Anesthesia
  Arms: Phenylephrine Group
Drug: Metaraminol — 200mcg Metaraminol after Spinal Anesthesia
  Arms: Metaraminol

SUMMARY:
It is a prospective clinical trial with random distribution that intends to investigate maternal and fetal effects of ephedrine, phenylephrine and metaraminol during cesarean delivery in patients with pre-eclampsia.

DETAILED DESCRIPTION:
Spinal anesthesia has become the main anesthetic technique for cesarean delivery due to avoidance of failed tracheal intubation risk, improvement of post-operative analgesia and promotion of early mother-neonate bonding. Spinal anesthesia should be safe and comfortable for mother and child when referring to the side effects, including hypotension. The choice of the best vasopressor in this context is approaching to a resolution, favoring phenylephrine use. However, studies on high-risk pregnancies are still required, such as uteroplacental insufficiency, preeclampsia and intra-uterine growth restriction cases. The purpose of this study is to compare the effects of the vasopressors ephedrine, phenylephrine and metaraminol on maternal cardiac output, uteroplacental and cerebral fetal blood flow in patients with preeclampsia under spinal anesthesia for cesarean delivery. Sixty pregnant patients will be recruited and randomly assigned to receive either ephedrine, phenylephrine or metaraminol, making a total of three groups with 20 patients each. Variables to be analyzed are uterine arterial pulsatility index, umbilical arterial pulsatility index, fetus middle cerebral artery pulsatility index, maternal cardiac output, maternal cardiac frequency, maternal mean arterial blood pressure and maternal peripheral vascular resistance. These variables will be recorded in three moments: before the spinal anesthesia with the patient in dorsal recumbent and left displacement of the uterus, after spinal anesthesia in dorsal recumbent and after vasopressor bolus. Averages will be calculated in these intervals and then compared to the alteration caused by spinal anesthesia and the return to basal levels after drug intervention.

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia patients
* After 34 weeks pregnant

Exclusion Criteria:

* Patients' refusal
* Obstetric Emergency
* Contraindications to spinal anesthesia
* Obesity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Middle cerebral artery pulsatility index changes before and after spinal anesthesia and vasopressor use. | One year
  The main purpose of this study is evaluate if one of related drugs (ephedrine, phenylephrine or metaraminol) is superior than others to keep the maternal cardiac output, uteroplacental and fetal cerebral bloodflow despite the hemodynamic changes that is peculiar after spinal anesthesia.
Maternal cardiac output changes after vasopressor (ephedrine, phenylephrine or metaraminol) use in pregnant patients under spinal anesthesia | One year
Uterine arterial pulsatility index changes before and after spinal anesthesia and vasopressor use. | One year
Umbilical arterial pulsatility index changes before an after spinal anesthesia and vasopressor use | One year

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bliacheriene, MD, Study Director — Instituto do Coracao
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil